CLINICAL TRIAL: NCT01179191
Title: A Multi-Center, Primary Care-Based, Open-Label Study to Assess the Success of Converting Opioid-Experienced Patients, With Chronic, Moderate to Severe Pain, to EMBEDA Using a Standardized Conversion Guide, and to Identify Behaviors Related to Prescription Opioid Abuse, Misuse, and Diversion
Brief Title: Conversion to Embeda With Rescue Trial
Acronym: ConvERT
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ALO-01-10-4003; B4541001
Record Dates: First submitted 2010-07-30; First posted 2010-08-11 (Estimated); Results first posted 2012-09-05 (Estimated); Last update posted 2012-10-11 (Estimated); Status verified 2012-10

CONDITIONS: Chronic Disease; Pain
Keywords: chronic pain; Embeda; opioid; moderate pain; severe pain; conversion; converting; switching; morphine; aberrant behavior; Pain (DT) + Chronic Disease (DT)
MeSH Terms: conditions — Chronic Disease; Pain; Chronic Pain | interventions — Morphine; Naltrexone; morphine, naltrexone combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- morphine sulfate and naltrexone hydrochloride (EMBEDA) (Experimental)
  Interventions: Drug: morphine sulfate and naltrexone hydrochloride (EMBEDA)

INTERVENTIONS:
Drug: morphine sulfate and naltrexone hydrochloride (EMBEDA) — Capsules in dose strengths ranging from 20 to 100 mg morphine sulfate with 0.8 to 4 mg of naltrexone hydrochloride taken either once or twice daily with a starting dose calculated using the total daily dose of the current opioid being converted from until a stable dose is achieved or six weeks which ever comes first.

SUMMARY:
The purpose of the research study is to find out if opioid dependent chronic pain patients who are judged by their physician to be eligible to change their current opioid medicine and to participate in this study can be successfully adjusted to a stable dose of EMBEDA (morphine sulfate and naltrexone hydrochloride). The study will also assess each patient's risk for prescription opioid abuse, misuse and diversion.

DETAILED DESCRIPTION:
The decision to terminate the trial was based on a lack of study drug supply. The decision was not based on any safety concerns. The termination letter was sent on 11March2011.

ELIGIBILITY:
Inclusion Criteria:

* Be able to read, speak and understand English
* Have chronic moderate to severe pain for at least 3 months
* Require around the clock opioid medication for the relief of pain
* Have been taking a daily opioid for at least 30 days prior to starting the study
* Be able to be safely switched to a different pain medication
* Be practicing acceptable birth control methods for female patients of childbearing potential
* Be willing to participate in the study and able to comply with study procedures

Exclusion Criteria:

* Be currently diagnosed with or participating in and/or seeking treatment for opioid and/or alcohol abuse
* Be allergic or intolerant to morphine, morphine salts, naltrexone or other opioids
* Be currently taking tramadol and/or extended release morphine products
* Have respiratory depression
* Have acute or severe bronchial asthma or severe chronic obstructive pulmonary disease
* Have migraines as your main source of pain
* Have any form of bowel obstruction
* Be pregnant or breast feeding
* Have had 2 or more surgeries for low back pain
* Be planning a major surgery during the study
* Be staying in a hospital or nursing home
* Be planning to have steroid injections for your chronic pain during the study
* Have a life expectancy of less than 2 months

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 684 (Actual)
Dates: Start 2010-08; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (164):
- United States (164):
  - Adamsville Family Medicine, Adamsville, Alabama
  - Office of David McLain, Birmingham, Alabama
  - Monte Sano Clinical Research, LLC, Huntsville, Alabama
  - Tennessee Valley Pain Consultants Properties, LLC, Huntsville, Alabama
  - Sunbelt Research Group, LLC, Mobile, Alabama
  - Office of Vaughn H. Mancha, Jr., PC, Montgomery, Alabama
  - Dedicated Clinical Research, Goodyear, Arizona
  - Dedicated Clinical Research, Inc, Phoenix, Arizona
  - Redpoint Research, Phoenix, Arizona
  - Anasazi Internal Medicine, PC, Phoenix, Arizona
  - Cochise Clinical Research, Sierra Vista, Arizona
  - Premiere Phamaceutical Research, LLC, Tempe, Arizona
  - Quality of Life Medical and Research Center, LLC, Tucson, Arizona
  - Ouachita Regional Pain Management, Hot Springs, Arkansas
  - NEA Baptist Clinic, Jonesboro, Arkansas
  - Hollis Family Medical Clinic, PLC, Paragould, Arkansas
  - CSI Clinical Trials, Costa Mesa, California
  - Global Wellness Medical Corporation, Foothill Ranch, California
  - Chrishard Medical Group, Inglewood, California
  - Triwest Research Associates LLC, La Mesa, California
  - Pacific Coast Pain Management Center, Laguna Hills, California
  - Valerius Medical Group and Research Center of Greater Long Beach, Inc., Long Beach, California
  - LA Pain & Wellness Institute, Los Angeles, California
  - Samaritan Center for Medical Research, Los Gatos, California
  - Newport Beach Clinical Research Associates, Inc., Newport Beach, California
  - Bayview Research Group, LLC, Paramount, California
  - Pasadena Rehabilitation Institute, Pasadena, California
  - Quality Control Research, Inc., Roseville, California
  - Northern California Research, Sacramento, California
  - Quality Control Research, Inc., Sacramento, California
  - Rancho Santa Fe Medical Group, Inc., San Marcos, California
  - Probe Clinical Research Corporation, Santa Ana, California
  - Trinity Clinical Trials, Santa Ana, California
  - Facility Medical Center, Upland, California
  - Bayview Research Group, LLC, Valley Village, California
  - Rocky Mountain Internal Medicine, PC, Aurora, Colorado
  - Clinicos, LLC, Colorado Springs, Colorado
  - Saint Luke's Medical Clinic, LLC, Fort Collins, Colorado
  - ProHealth Physicians PC, Manchester, Connecticut
  - Milford Physician Services, PC, Milford, Connecticut
  - Orthopedic Research Institute, LLC, Boynton Beach, Florida
  - Florida Research & Testing, LLC, Clearwater, Florida
  - Omega Research Consultants, LLC, DeBary, Florida
  - West Florida Medical Associate, PA, Dunnellon, Florida
  - International Research Associates, LLC, Hialeah, Florida
  - Palm Springs Research Institute, Inc, Hialeah, Florida
  - FPA Clinical Research, LLC, Kissimmee, Florida
  - Clinical Research of Central Florida, Inc., Lakeland, Florida
  - Community Research Foundation, Inc., Miami, Florida
  - New Horizon Research Center, Inc., Miami, Florida
  - NextPhase Clinical Trials, Inc., Miami Beach, Florida
  - Harmony Clinical Research, Inc., North Miami Beach, Florida
  - Office of Laszlo J. Mate, MD, PA, North Palm Beach, Florida
  - Office of Richard E. Promin, MD, PA, Ocala, Florida
  - Advent Clinical Research Centers, Inc., Pinellas Park, Florida
  - Pain Management Strategies, Inc., Pompano Beach, Florida
  - Sarasota Pain Medicine Research, LLC, Sarasota, Florida
  - Stedman Clinical Trials, LLC, Tampa, Florida
  - Clinical Research Center, LLC, Wellington, Florida
  - Perimeter Institute for Clinical Research, Inc., Atlanta, Georgia
  - Medical Research and Health Education Foundation, Inc., Columbus, Georgia
  - Ialum Clinical Research, LLC, Decatur, Georgia
  - Ialum Clinical Research, LLC, Stone Mountain, Georgia
  - Herman Clinical Research, LLC, Suwanee, Georgia
  - Centers for Pain Management, Tifton, Georgia
  - Chicago Clinical Research Institute Inc., Chicago, Illinois
  - Creve Coeur Family Practice, Creve Coeur, Illinois
  - Office of Rebecca Knight, MD, Peoria, Illinois
  - Josephson Wallack Munshower Neurology P.C., Indianapolis, Indiana
  - Laporte County Institute for Clinical Research Inc., Michigan City, Indiana
  - McKinley Research, LLC, Mishawaka, Indiana
  - Accelovance, Inc., South Bend, Indiana
  - Des Moines Orthopaedic Surgeons, PC, West Des Moines, Iowa
  - The Pain Treatment Center of the Bluegrass, Lexington, Kentucky
  - Healing Options, Louisville, Kentucky
  - Four Rivers Clinical Research, Inc., Paducah, Kentucky
  - Lakewood Family Practice, Russell Springs, Kentucky
  - Diseasebusters, LLC, College Park, Maryland
  - Office of Steven C. Miller, MD, Pikesville, Maryland
  - Beacon Clinical Research, LLC, Brockton, Massachusetts
  - Ronald J. Rapoport, MD, PC, Fall River, Massachusetts
  - Boston Paincare Center, Inc., Waltham, Massachusetts
  - Clarkston Medical Group, PC, Clarkston, Michigan
  - Apex Medical Research, AMR, Inc., Flint, Michigan
  - East Michigan Medical Associates, Flint, Michigan
  - PCM Medical Services, PC, Lansing, Michigan
  - Remedica LLC, Rochester, Michigan
  - Michigan Lifestyle Change and Health Center, PC, Sterling, Michigan
  - MAPS Applied Research Center, Inc., Edina, Minnesota
  - MAPS Applied Research Center, Inc., Shakopee, Minnesota
  - Anesthesia and Pain Control Services, Biloxi, Mississippi
  - CRC of Jackson, LLC, Jackson, Mississippi
  - Midsouth Anesthesia Consultants, PLLC, Southhaven, Mississippi
  - Patterson Medical Clinic, Inc., Florissant, Missouri
  - Quality Clinical Research Inc., Florissant, Missouri
  - Primary Care Medicine, PC, Jefferson City, Missouri
  - The Reiter Foundation, Inc., Anaconda, Montana
  - Medical Pain Relief Clinic, Omaha, Nebraska
  - Omaha Clinical Research, PC, Omaha, Nebraska
  - Atco Medical Associates, PC, Atco, New Jersey
  - Office of John V. Bernard, MD, Belvidere, New Jersey
  - Central Jersey Medical Research Center, Inc., Elizabeth, New Jersey
  - Center for Pain Management, Hackensack, New Jersey
  - Advocare Heights Primary Care, Haddon Heights, New Jersey
  - NJ Heart, LLC, Linden, New Jersey
  - Spine and Pain Centers, PA, Shrewsbury, New Jersey
  - Premier Research, Inc., Trenton, New Jersey
  - Adirondack Medical Research Center, Glens Falls, New York
  - Long Island Gastrointestinal Research Group LLP, Great Neck, New York
  - Drug Trials America, Inc., Hartsdale, New York
  - Office of Roger Kasendorf, DO, Long Beach, New York
  - Family Health Medical Services PLLC, Mayville, New York
  - New York Spine & Wellness Center, North Syracuse, New York
  - North American Partners in Pain Management, LLP, Valley Stream, New York
  - Carolina Clinical Research and Consulting, LLC, Asheboro, North Carolina
  - Joint and Muscle Research Institute, Inc., Charlotte, North Carolina
  - Catawba Valley Internal Medicine, Hickory, North Carolina
  - Profen Research Network at ECMA, Jacksonville, North Carolina
  - The Center For Clinical Research, LLC, Winston-Salem, North Carolina
  - Medical Frontiers, LLC, Carlisle, Ohio
  - Valley Medical Research, Centerville, Ohio
  - Hightop Medical Research Center, Cincinnati, Ohio
  - Sentral Clinical Research Services, Cincinnati, Ohio
  - Delaware Smith Clinic Research, Delaware, Ohio
  - Medical Frontiers, LLC, Franklin, Ohio
  - Jeffrey J. Haggenjos, DO, Inc., New Lexington, Ohio
  - Whole Family Medical Care LLC, Perrysburg, Ohio
  - Office of Jocelyn F. Shimek, DO, Salem, Ohio
  - Office of James Lassiter, Tiffin, Ohio
  - Health Research Institute, LLC, Oklahoma City, Oklahoma
  - Office of Siavash Nael, MD, Inc., Oklahoma City, Oklahoma
  - Associates of Medicine/John D. Williams, MD, PLLC, Stillwater, Oklahoma
  - Portland Rheumatology Clinic, LLC, Lake Oswego, Oregon
  - Office of Joseph E. Yankee, DO, PC, Milwaukie, Oregon
  - Pennsylvania Pain Specialists, PC, Allentown, Pennsylvania
  - Ware Medical Associates, PC, Aston Mills, Pennsylvania
  - Altoona Center for Clinical Research, PC, Duncansville, Pennsylvania
  - Kandra, Fierer, Kuskin Associates, Ltd., Harrisburg, Pennsylvania
  - Onuorah Umeh, M.D. P.C, Philadelphia, Pennsylvania
  - Founders Research Corporation, Philadelphia, Pennsylvania
  - Progressive Pain Solutions, LLC, Wind Gap, Pennsylvania
  - Hartwell Research Group, LLC, Anderson, South Carolina
  - Low Country Rheumatology, PA, Charleston, South Carolina
  - Pharmacorp Clinical Trials, Inc., Charleston, South Carolina
  - Internal Medicine of Greer Research LLC, Greer, South Carolina
  - Clinical Research Authority, LLC, Murrells Inlet, South Carolina
  - Trident Institute of Medical Research, LLC, North Charleston, South Carolina
  - Low Country Pain Center, LLC, Orangeburg, South Carolina
  - Brown Clinic, PLLP, Watertown, South Dakota
  - Chattanooga Medical Research, LLC, Chattanooga, Tennessee
  - Comprehensive Pain Specialists, Hendersonville, Tennessee
  - Corsicana Medical Research, PLLC, Corsicana, Texas
  - DCT - Genesis Neighborhood Research, LLC, Dallas, Texas
  - Southwest Urgent Care Center, El Paso, Texas
  - Westbury Medical Clinic, Houston, Texas
  - Accurate Clinical Research, Inc., Houston, Texas
  - Medstar Clinical Research, Houston, Texas
  - Texas Medical Research Associates, LLC, San Antonio, Texas
  - Hillcrest Family Health Center, Division of Clinical Research, Waco, Texas
  - Hillcrest Family Health Center, Waco, Texas
  - Progressive Clinical Research, LLC, Bountiful, Utah
  - Sentara Medical Group, NDC Medical Center, Norfolk, Virginia
  - Washington Center for Pain Management PLLC, Edmonds, Washington
  - Pain Care, PLLC, Huntington, West Virginia

REFERENCES:
- [Derived] Setnik B, Roland CL, Pixton GC, Sommerville KW. Prescription opioid abuse and misuse: gap between primary-care investigator assessment and actual extent of these behaviors among patients with chronic pain. Postgrad Med. 2017 Jan;129(1):5-11. doi: 10.1080/00325481.2017.1245585. Epub 2016 Oct 26. PMID 27782769
- [Derived] Setnik B, Roland CL, Sommerville KW, Pixton GC, Berke R, Calkins A, Goli V. A multicenter, primary-care-based, open-label study to assess the success of converting opioid-experienced patients with chronic moderate-to-severe pain to morphine sulfate and naltrexone hydrochloride extended-release capsules using a standardized conversion guide. J Pain Res. 2015 Jul 8;8:347-60. doi: 10.2147/JPR.S82395. eCollection 2015. PMID 26185466
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=ALO-01-10-4003&StudyName=Conversion%20to%20Embeda%20With%20Rescue%20Trial

RESULTS

PARTICIPANT FLOW:
Groups:
- EMBEDA: EMBEDA (morphine sulfate/naltrexone hydrochloride) extended-release capsules orally prescribed according to usual clinical practice using a standardized conversion guide. Treatment included titration phase (up to 6 weeks) followed by maintenance phase (8 weeks).
Period: Titration Phase (up to 6 Weeks)
Arm/Group | EMBEDA
Started | 684
Completed | 351
Not Completed | 333
Not completed — Adverse Event | 47
Not completed — Lost to Follow-up | 19
Not completed — Physician Decision | 30
Not completed — Withdrawal by Subject | 162
Not completed — Participant did not reach stable dose | 13
Not completed — Other | 62
Period: Maintenance Phase (8 Weeks)
Arm/Group | EMBEDA
Started | 351
Completed | 234
Not Completed | 117
Not completed — Adverse Event | 10
Not completed — Lost to Follow-up | 9
Not completed — Physician Decision | 3
Not completed — Withdrawal by Subject | 29
Not completed — Other | 66

BASELINE CHARACTERISTICS:
Arm/Group | EMBEDA
Number analyzed (Participants) | 684
Age Continuous [Mean (Standard Deviation); unit: Years] | 51.77 (12.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 378
  Male | 306
Brief Pain Inventory (BPI) [Mean (Standard Deviation); unit: Units on a scale] — BPI:11-item questionnaire,4 questions:pain intensity(worst,least,average,relief),7questions:pain impact on daily functions(general activity,mood,walking ability,normal work,relations with others,sleep,life enjoyment).Each question range=0-10(0%-100% for relief),higher score=more pain/relief/interference.'n'=participants evaluated for each subscale.
  Units on a scale
    Average Pain (n = 636) | 6.27 (1.79)
    Worst Pain (n = 636) | 7.95 (1.64)
    Least Pain (n = 642) | 4.63 (2.27)
    Relief (n = 639) | 53.36 (22.72)
    General Activity (n = 643) | 7.01 (2.33)
    Mood (n = 642) | 6.31 (2.73)
    Walking Ability (n = 641) | 6.48 (2.78)
    Normal Work (n = 637) | 7.21 (2.48)
    Relationships with Others (n = 644) | 5.41 (3.08)
    Sleep (n = 642) | 6.80 (2.74)
    Enjoyment of Life (n = 640) | 7.03 (2.64)
Investigator(Ir) Compared to Participant(Pa)-Derived Risk Level Assessment of Misuse,Abuse,Diversion [Number; unit: Participants] — Number of participants at Ir-assessed risk level compared to Pa-derived risk level (low,moderate[mod] or high) for opioid misuse,abuse,diversion. An exploratory scoring algorithm applied to results of Participant's Experience and Concerns Questionnaire to get Pa-derived risk levels. Pa evaluable=683. 'n'=Pa evaluated for each assessed risk level.
  Participants
    Abuse: Low(Ir)/ Low(Pa) (n= 6) | 6
    Abuse: Low(Ir)/ Moderate (Mod)(Pa) (n= 6) | 0
    Abuse: Low(Ir)/ High(Pa) (n= 6) | 0
    Abuse: Mod(Ir)/ Low(Pa) (n= 1) | 1
    Abuse: Mod(Ir)/ Mod(Pa) (n= 1) | 0
    Abuse: Mod(Ir)/ High(Pa) (n= 1) | 0
    Abuse: High(Ir)/ Low(Pa) (n= 1) | 0
    Abuse: High(Ir)/ Mod(Pa) (n= 1) | 1
    Abuse: High(Ir)/ High(Pa) (n= 1) | 0
    Misuse General: Low(Ir)/ Low(Pa) (n= 127) | 118
    Misuse General: Low(Ir)/ Mod(Pa) (n= 127) | 9
    Misuse General: Low(Ir)/ High(Pa) (n= 127) | 0
    Misuse General: Mod(Ir)/ Low(Pa) (n= 24) | 22
    Misuse General: Mod(Ir)/ Mod(Pa) (n= 24) | 2
    Misuse General: Mod(Ir)/ High(Pa) (n= 24) | 0
    Misuse General: High(Ir)/ Low(Pa) (n= 3) | 2
    Misuse General: High(Ir)/ Mod(Pa) (n= 3) | 1
    Misuse General: High(Ir)/ High(Pa) (n= 3) | 0
    Misuse Pseudoaddiction: Low(Ir)/ Low(Pa) (n= 227) | 208
    Misuse Pseudoaddiction: Low(Ir)/ Mod(Pa) (n= 227) | 18
    Misuse Pseudoaddiction: Low(Ir)/ High(Pa) (n= 227) | 1
    Misuse Pseudoaddiction: Mod(Ir)/ Low(Pa) (n= 42) | 38
    Misuse Pseudoaddiction: Mod(Ir)/ Mod(Pa) (n= 42) | 3
    Misuse Pseudoaddiction: Mod(Ir)/ High(Pa) (n= 42) | 1
    Misuse Pseudoaddiction: High(Ir)/ Low(Pa) (n= 5) | 3
    Misuse Pseudoaddiction: High(Ir)/ Mod(Pa) (n= 5) | 1
    Misuse Pseudoaddiction: High(Ir)/ High(Pa) (n= 5) | 1
    Misuse Total: Low(Ir)/ Low(Pa) (n= 295) | 245
    Misuse Total: Low(Ir)/ Mod(Pa) (n= 295) | 49
    Misuse Total: Low(Ir)/ High(Pa) (n= 295) | 1
    Misuse Total: Mod(Ir)/ Low(Pa) (n= 56) | 40
    Misuse Total: Mod(Ir)/ Mod(Pa) (n= 56) | 14
    Misuse Total: Mod(Ir)/ High(Pa) (n= 56) | 2
    Misuse Total: High(Ir)/ Low(Pa) (n= 6) | 3
    Misuse Total: High(Ir)/ Mod(Pa) (n= 6) | 2
    Misuse Total: High(Ir)/ High(Pa) (n= 6) | 1
    Diversion: Low (Ir)/ Low (Pa) (n= 487) | 467
    Diversion: Low (Ir)/ Mod (Pa) (n= 487) | 10
    Diversion: Low (Ir)/ High (Pa) (n= 487) | 10
    Diversion: Mod (Ir)/ Low (Pa) (n= 22) | 19
    Diversion: Mod (Ir)/ Mod (Pa) (n= 22) | 2
    Diversion: Mod (Ir)/ High (Pa) (n= 22) | 1
    Diversion: High (Ir)/ Low (Pa) (n= 5) | 3
    Diversion: High (Ir)/ Mod (Pa) (n= 5) | 0
    Diversion: High (Ir)/ High (Pa) (n= 5) | 2
Number of Participants Reporting Concerns With Prescription Opioid (Op) Misuse, Abuse or Diversion [Number; unit: Participants] — Participant experience and concerns with prescription opioids questionnaire consisted of multiple choice questions and numeric rating scale(NRS);range=0(not at all) to 10 (extremely worried);used to assess current concerns, past behaviors related to opioid misuse, abuse, diversion.n=Pa evaluable for given question. Pa may choose more than 1 reason.
  Participants
    Worried getting addicted or hooked to Op:0(n=537) | 171
    Worried getting addicted or hooked to Op:1(n=537) | 47
    Worried getting addicted or hooked to Op:2(n=537) | 53
    Worried getting addicted or hooked to Op:3(n=537) | 47
    Worried getting addicted or hooked to Op:4(n=537) | 30
    Worried getting addicted or hooked to Op:5(n=537) | 53
    Worried getting addicted or hooked to Op:6(n=537) | 28
    Worried getting addicted or hooked to Op:7(n=537) | 33
    Worried getting addicted or hooked to Op:8(n=537) | 31
    Worried getting addicted or hooked to Op:9(n=537) | 11
    Worried getting addicted or hooked to Op:10(n=537) | 33
    Worried about hard time to stop Op:0(n=537) | 138
    Worried about hard time to stop Op:1(n=537) | 50
    Worried about hard time to stop Op:2(n=537) | 67
    Worried about hard time to stop Op:3(n=537) | 45
    Worried about hard time to stop Op:4(n=537) | 20
    Worried about hard time to stop Op:5(n=537) | 54
    Worried about hard time to stop Op:6(n=537) | 26
    Worried about hard time to stop Op:7(n=537) | 39
    Worried about hard time to stop Op:8(n=537) | 35
    Worried about hard time to stop Op:9(n=537) | 27
    Worried about hard time to stop Op:10(n=537) | 36
    Chewed/crushed Op:tried once/twice(n=534) | 31
    Chewed/crushed Op:few times a year(n=534) | 5
    Chewed/crushed Op:few times a month(n=534) | 10
    Chewed/crushed Op:few times a week(n=534) | 7
    Chewed/crushed Op:daily(n=534) | 5
    Chewed/crushed Op:never(n=534) | 476
    Reason(Rn)to chew/crush Op:treat pain better(n=71) | 35
    Rn to chew/crush Op:treat new pain(n=71) | 4
    Rn to chew/crush Op:sleep better/relax(n=71) | 14
    Rn to chew/crush Op:help swallow drug(n=71) | 16
    Rn to chew/crush Op:feel pleasant/high(n=71) | 3
    Rn to chew/crush Op:feel less depressed (n=71) | 6
    Rn to chew/crush Op:feel talkative/outgoing(n=71) | 2
    Rn to chew/crush Op:other(n=71) | 29
    More Op than prescribed:tried once/twice(n=530) | 75
    More Op than prescribed:few times a year(n=530) | 46
    More Op than prescribed:few times a month(n=530) | 116
    More Op than prescribed:few times a week(n=530) | 58
    More Op than prescribed:daily(n=530) | 23
    More Op than prescribed:never(n=530) | 212
    Rn for more Op use:treat pain better(n=315) | 274
    Rn for more Op use:treat new pain(n=315) | 42
    Rn for more Op use:sleep better/relax(n=315) | 48
    Rn for more Op use:feel pleasant/high(n=315) | 3
    Rn for more Op use:feel less depressed (n=315) | 16
    Rn for more Op use:feel talkative/outgoing(n=315) | 3
    Rn for more Op use: other(n=315) | 44
    Snort,smoke,inject(inj) Op:once/twice(n=533) | 7
    Snort,smoke,inj Op: few times a year(n=533) | 0
    Snort,smoke,inj Op:few times a month(n=533) | 2
    Snort,smoke,inj Op:few times a week(n=533) | 0
    Snort,smoke,inj Op:daily(n=533) | 1
    Snort,smoke,inj Op:never(n=533) | 523
    Rn-snort,smoke,inj:treat pain better(n=37) | 10
    Rn-snort,smoke,inj:treat new pain (n=37) | 1
    Rn-snort,smoke,inj:sleep better/relax(n=37) | 2
    Rn-snort,smoke,inj:feel pleasant/high(n=37) | 2
    Rn-snort,smoke,inj:feel less depressed (n=37) | 2
    Rn-snort,smoke,inj:feel talkative/outgoing(n=37) | 2
    Rn-snort,smoke,inj:other(n=37) | 28
    Alcohol(Alc)use when on Op:tried once/twice(n=534) | 32
    Alc use when on Op:few times a year(n=534) | 50
    Alc use when on Op:few times a month(n=534) | 35
    Alc use when on Op:few times a week(n=534) | 19
    Alc use when on Op:daily(n=534) | 7
    Alc use when on Op:never(n=534) | 391
    Rn-Alc when on Op:treat pain better(n=170) | 10
    Rn-Alc when on Op:treat new pain(n=170) | 1
    Rn-Alc when on Op:sleep better/relax(n=170) | 21
    Rn-Alc when on Op:enjoy occasional drink(n=170 | 91
    Rn-Alc when on Op:feel pleasant/high(n=170) | 3
    Rn-Alc when on Op:feel less depressed(n=170) | 4
    Rn-Alc when on Op:feel talkative/outgoing(n=170) | 2
    Rn-Alc when on Op:other(n=170) | 65
    More than 1 doctor (Dr) for Op:once/twice(n=529) | 26
    More than 1 Dr for Op:sometime(n=529) | 12
    More than 1 Dr for Op:often(n=529) | 3
    More than 1 Dr for Op:never(n=529) | 488
    Rn- more than 1 Dr:treat pain better(n=61) | 26
    Rn- more than 1 Dr: prevent withdrawal(n=61) | 6
    Rn- more than 1 Dr:afraid to ask for more(n=61) | 12
    Rn- more than 1 Dr:feel pleasant/high (n=61) | 1
    Rn- more than 1 Dr:Dr didn't prescribed more(n=61) | 11
    Rn- more than (>) 1 Dr:other(n=61) | 24
    Gave Op to sick/in pain:yes (n=526) | 35
    Gave Op to sick/in pain:yes,once(n=35) | 5
    Gave Op to sick/in pain:yes, 2-5times(n=35) | 24
    Gave Op to sick/in pain:yes,6-10times(n=35) | 3
    Gave Op to sick/in pain:yes, >10 times(n=35) | 3
    Gave Op to sick/in pain:no(n=526) | 491
    Got Op from someone other than a doctor:yes(n=537) | 43
    Got Op from someone other than a doctor:no(n=537) | 494
    Keeps Op hidden or locked:yes(n=535) | 373
    Keeps Op hidden or locked:no(n=535) | 162
    Suspected someone taking Op:yes(n=535) | 71
    Suspected someone taking Op:yes,once(n=70) | 30
    Suspected someone taking Op:yes,few times(n=70) | 29
    Suspected someone taking Op:yes,sometimes (n=70) | 8
    Suspected someone taking Op:yes,all times (n=70) | 3
    Suspected someone taking Op:no(n=535) | 464

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Stable Dose of EMBEDA Within 6 Weeks Titration Phase
Description: A dose was considered to be stable dose if it met all of the following criteria: dose was taken for at least 48 hours; investigator deemed the balance between an acceptable level of analgesia and/or function and tolerance of side effects had been achieved; and rescue medication use less than or equal to 2 doses per day.
Time Frame: Baseline through Week 6
Population: Safety population included all participants who completed the first study visit and filled a prescription for EMBEDA.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | EMBEDA
Number analyzed (Participants) | 684
Percentage of participants | 51.3 [47.5 to 55.1]

2. Primary Outcome: Percentage of Participants Achieving Stable Dose of EMBEDA Within 6 Weeks Titration Phase Stratified by Prior Opioid Therapy
Description: as for outcome 1
Time Frame: Baseline through Week 6
Population: Safety population included all participants who completed the first study visit and filled a prescription for EMBEDA. Participants were stratified based on prior opioid therapy. The 'n' is signifying those participants who were evaluated for this measure for each of the prior medication received.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | EMBEDA
Number analyzed (Participants) | 684
Percentage of participants
  Transdermal Fentanyl (n= 77) | 54.5 [42.8 to 65.9]
  Immediate-release (IR) Hydrocodone (n= 164) | 60.4 [52.4 to 67.9]
  IR Hydromorphone (n= 22) | 63.6 [40.7 to 82.8]
  IR Oxycodone (n= 160) | 48.1 [40.2 to 56.2]
  IR Morphine (n= 53) | 62.3 [47.9 to 75.2]
  Methadone (n= 64) | 40.6 [28.5 to 53.6]
  Extended-release (ER) Oxycodone (n= 107) | 42.1 [32.6 to 52.0]
  ER Oxymorphone (n= 25) | 56.0 [34.9 to 75.6]
  Excluded Opioid/ Unclassified (n= 12) | 8.3 [0.2 to 38.5]

3. Secondary Outcome: Duration to Titrate Participants to Stable Dose
Description: as for outcome 1
Time Frame: Baseline through Week 6
Population: Safety population included all participants who completed the first study visit and filled a prescription for EMBEDA. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | EMBEDA
Number analyzed (Participants) | 351
Days | 20.0 (8.94)

4. Secondary Outcome: Duration to Titrate Participants to Stable Dose Stratified by Prior Opioid Therapy
Description: as for outcome 1
Time Frame: Baseline through Week 6
Population: Safety population. Participants were stratified based on prior opioid therapy. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure. 'n' signifies those participants who were evaluated for this measure for each of the prior medication received.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | EMBEDA
Number analyzed (Participants) | 351
Days
  Transdermal Fentanyl (n= 42) | 17.8 (5.96)
  IR Hydrocodone (n= 99) | 20.7 (9.13)
  IR Hydromorphone (n= 14) | 24.3 (12.55)
  IR Oxycodone (n= 77) | 19.6 (8.35)
  IR Morphine (n= 33) | 18.8 (7.82)
  Methadone (n= 26) | 21.0 (8.70)
  ER Oxycodone (n= 45) | 20.3 (10.55)
  ER Oxymorphone (n= 14) | 19.8 (10.71)
  Excluded Opioid/ Unclassified (n= 1) | 7.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.

5. Secondary Outcome: Number of Titration Steps to Achieve Stable Dose
Description: as for outcome 1
Time Frame: Baseline through Week 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: titration steps
Arm/Group | EMBEDA
Number analyzed (Participants) | 351
titration steps | 2.4 (1.37)

6. Secondary Outcome: Number of Titration Steps to Achieve Stable Dose Stratified by Prior Opioid Therapy
Description: as for outcome 1
Time Frame: Baseline through Week 6
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: titration steps
Arm/Group | EMBEDA
Number analyzed (Participants) | 351
titration steps
  Transdermal Fentanyl (n= 42) | 2.0 (0.98)
  IR Hydrocodone (n= 99) | 2.6 (1.41)
  IR Hydromorphone (n= 14) | 2.6 (1.28)
  IR Oxycodone (n= 77) | 2.3 (1.40)
  IR Morphine (n= 33) | 2.3 (1.28)
  Methadone (n= 26) | 2.7 (1.52)
  ER Oxycodone (n= 45) | 2.4 (1.50)
  ER Oxymorphone (n= 14) | 2.5 (1.45)
  Excluded Opioid/ Unclassified (n= 1) | 1.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.

7. Secondary Outcome: Percentage of Participants With Rescue Medications Usage During Titration
Description: Rescue pain medications were used for supplemental analgesia for breakthrough pain during titration phase. Morphine sulfate IR tablet (less than 20 percent of the total daily dose of EMBEDA per IR dose), ibuprofen (up to 400 milligram (mg)/dose; not to exceed 1200 mg/day), and acetaminophen (up to 1000 mg/dose, not to exceed 4000 mg/day) were used as rescue medications.
Time Frame: Baseline through Week 6
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | EMBEDA
Number analyzed (Participants) | 650
Percentage of participants | 79.8

8. Secondary Outcome: Change From Baseline in Brief Pain Inventory (BPI) at Visit 3 (First Visit After Successful Titration)
Description: BPI is an 11-item self-report questionnaire: consist of 4 questions that assess pain intensity (worst, least, average, relief) and 7 questions that assess impact of pain on daily functions (general activity, mood, walking ability, normal work, relations with other people, sleep, enjoyment of life). Each question answered on a scale range:0-10 (0%-100% for relief), '0=No pain/no relief/no interference and 10=Pain as bad as you can imagine/complete relief/ complete interference'.Measure can be scored by item, with lower scores being indicative of less pain or pain interference.
Time Frame: Baseline, Visit 3 (up to Week 6)
Population: Safety population included all participants who completed the first study visit and filled a prescription for EMBEDA. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure. The 'n' is signifying those participants who were evaluated for the respective subscale.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | EMBEDA
Number analyzed (Participants) | 322
Units on a scale
  Change at Visit 3 (Average Pain) (n=313) | -2.23 (2.13)
  Change at Visit 3 (Worst Pain) (n=313) | -2.41 (2.49)
  Change at Visit 3 (Least Pain) (n=321) | -1.81 (2.33)
  Change at Visit 3 (Relief) (n=0) | NA (NA) — Data for this component of BPI was not summarized as analysis plan focused on average, worst and least pain components of the BPI.
  Change at Visit 3 (General Activity) (n=0) | NA (NA) — Data for this component of BPI was not summarized as analysis plan focused on average, worst and least pain components of the BPI.
  Change at Visit 3 (Mood) (n=0) | NA (NA) — Data for this component of BPI was not summarized as analysis plan focused on average, worst and least pain components of the BPI.
  Change at Visit 3 (Walking Ability) (n=0) | NA (NA) — Data for this component of BPI was not summarized as analysis plan focused on average, worst and least pain components of the BPI.
  Change at Visit 3 (Normal Work) (n=0) | NA (NA) — Data for this component of BPI was not summarized as analysis plan focused on average, worst and least pain components of the BPI.
  Change at Visit 3(Relationships with Others) (n=0) | NA (NA) — Data for this component of BPI was not summarized as analysis plan focused on average, worst and least pain components of the BPI.
  Change at Visit 3 (Sleep) (n=0) | NA (NA) — Data for this component of BPI was not summarized as analysis plan focused on average, worst and least pain components of the BPI.
  Change at Visit 3 (Enjoyment of Life) (n=0) | NA (NA) — Data for this component of BPI was not summarized as analysis plan focused on average, worst and least pain components of the BPI.

9. Secondary Outcome: Investigator's Level of Satisfaction With the EMBEDA Conversion Guide
Description: The conversion assessment survey is a brief questionnaire using multiple choice options and numeric rating scale (NRS) with specified anchored responses ranging on a scale from 0-10 (0 = very dissatisfied, 5 = neutral, and 10=very satisfied) to assess the Investigator's level of satisfaction with the EMBEDA Conversion Guide.
Time Frame: Week 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | EMBEDA
Number analyzed (Participants) | 349
Units on a Scale | 8.1 (2.11)

10. Other Pre Specified Outcome: Number of Participants With Aberrant Behaviors
Description: Current Opioid Misuse Measure (COMM) is a 17-item self-administered test used to monitor aberrant behavior in participants on opioid therapy. Aberrant behaviors assessed using a 5-point scale [0 = 'never' and 4 = 'very often']. Score range 0-68. Scores greater than or equal to 9 indicated the presence of aberrant behaviors.
Time Frame: Day 5
Population: Safety population included all participants who completed the first study visit and filled a prescription for EMBEDA.
Measure: Number; unit: Participants
Arm/Group | EMBEDA
Number analyzed (Participants) | 684
Participants | 217

11. Other Pre Specified Outcome: Number of Participants With Abnormal Urine Drug Test Results
Description: Urine samples collected were screened using immunoassay techniques for the following types of drugs: opioids, barbiturates, benzodiazepines, amphetamines, ecstasy [3, 4-methylenedioxyamphetamine (MDMA)], cocaine, phencyclidine (PCP) and marijuana [tetrahydrocannabinol (THC)]. Quantitative, confirmatory urine drug testing was performed for positive results using gas chromatography or high-pressure liquid chromatography, for the following analytes: morphine, oxycodone, oxymorphone, hydrocodone, hydromorphone, fentanyl, methadone, benzodiazepines, amphetamines, cocaine, THC, PCP, and MDMA.
Time Frame: Baseline, Visit 3 (up to Week 6)
Population: Safety population included all participants who completed the first study visit and filled a prescription for EMBEDA. Here, the 'n' is signifying those participants who were evaluable for this measure at the specified time point for this arm group.
Measure: Number; unit: Participants
Arm/Group | EMBEDA
Number analyzed (Participants) | 684
Participants
  Baseline (n= 684) | 160
  Visit 3 (n= 351) | 101

12. Other Pre Specified Outcome: Number of Participants With Urine Drug Test Results Positive for Unaccounted Opioids
Description: Urine samples collected were screened using immunoassay techniques for the following types of drugs: opioids, barbiturates, benzodiazepines, amphetamines, ecstasy (3, 4-MDMA), cocaine, PCP and marijuana (THC). Quantitative, confirmatory urine drug testing was performed for positive results using gas chromatography or high-pressure liquid chromatography, for the following analytes: morphine, oxycodone, oxymorphone, hydrocodone, hydromorphone, fentanyl, methadone, benzodiazepines, amphetamines, cocaine, THC, PCP, and MDMA.
Time Frame: Visit 3 (up to Week 6)
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | EMBEDA
Number analyzed (Participants) | 351
Participants | 85

13. Other Pre Specified Outcome: Number of Participants With Urine Drug Test Results Positive for Illicit Substances
Description: Urine samples collected were screened using immunoassay techniques for following types of drugs:opioids,barbiturates,benzodiazepines,amphetamines,ecstasy(3,4MDMA),cocaine,PCP,marijuana (THC).Quantitative, confirmatory urine drug testing performed for positive results using gas chromatography or high-pressure liquid chromatography for following analytes: morphine,oxycodone,oxymorphone,hydrocodone,hydromorphone,fentanyl,methadone,benzodiazepines,amphetamines,cocaine,THC,PCP,MDMA. Illicit substances were drugs of categories:marijuana (THC) metabolite,cocaine metabolite,PCP,amphetamine.
Time Frame: Baseline, Visit 3 (up to Week 6)
Population: as for outcome 11
Measure: Number; unit: Participants
Arm/Group | EMBEDA
Number analyzed (Participants) | 684
Participants
  Baseline (n= 684) | 51
  Visit 3 (n= 351) | 24

14. Other Pre Specified Outcome: Number of Participants With Greater Than or Equal to One Urine Drug Test Results Negative for Expected Opioid
Description: as for outcome 12
Time Frame: Baseline, Visit 3 (up to Week 6)
Population: as for outcome 11
Measure: Number; unit: Participants
Arm/Group | EMBEDA
Number analyzed (Participants) | 684
Participants
  Baseline (n= 684) | 122
  Visit 3 (n= 351) | 11

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | EMBEDA
Serious Adverse Events (participants affected / at risk) | 24/684
Other Adverse Events (participants affected / at risk) | 331/684
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EMBEDA (N=684)
Angina unstable (Cardiac disorders) | 1
Dyspnoea (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Right ventricular hypertrophy (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Hyperglycaemia (Endocrine disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Diverticulitis (Gastrointestinal disorders) | 1
Gastroenteritis (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 1
Sudden death (General disorders) | 1
Hepatitis acute (Hepatobiliary disorders) | 1
Skin infection (Infections and infestations) | 1
Radius fracture (Injury, poisoning and procedural complications) | 1
Electrocardiogram t wave inversion (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Gout (Metabolism and nutrition disorders) | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1
Carotid artery disease (Nervous system disorders) | 1
Convulsion (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Dyskinesia (Nervous system disorders) | 1
Transient ishaemic attack (Nervous system disorders) | 1
Drug abuse (Psychiatric disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EMBEDA (N=684)
Anaemia (Blood and lymphatic system disorders) | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Bradycardia (Cardiac disorders) | 1
Dyspnoea (Cardiac disorders) | 5
Oedema peripheral (Cardiac disorders) | 3
Palpitations (Cardiac disorders) | 1
Syncope (Cardiac disorders) | 2
Tachycardia (Cardiac disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Diabetes mellitus (Endocrine disorders) | 1
Blindness transient (Eye disorders) | 1
Cataract (Eye disorders) | 1
Diplopia (Eye disorders) | 1
Eye pain (Eye disorders) | 1
Metamorphopsia (Eye disorders) | 1
Scleral haemorrhage (Eye disorders) | 1
Vision blurred (Eye disorders) | 6
Abdominal discomfort (Gastrointestinal disorders) | 3
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 10
Breath odour (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 74
Crohn's disease (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 8
Dry mouth (Gastrointestinal disorders) | 11
Dysgeusia (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 4
Enteritis infectious (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Food poisoning (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastroenteritis viral (Gastrointestinal disorders) | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 55
Painful defaecation (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Tooth disorder (Gastrointestinal disorders) | 1
Tooth infection (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 33
Adverse drug reaction (General disorders) | 4
Adverse event (General disorders) | 1
Asthenia (General disorders) | 1
Burning sensation (General disorders) | 2
Chest discomfort (General disorders) | 2
Chest pain (General disorders) | 4
Chills (General disorders) | 5
Drug intolerance (General disorders) | 1
Drug withdrawal syndrome (General disorders) | 1
Face oedema (General disorders) | 1
Fatigue (General disorders) | 20
Feeling abnormal (General disorders) | 1
Feeling of body temperature change (General disorders) | 1
Flushing (General disorders) | 2
Gait disturbance (General disorders) | 1
Hot flush (General disorders) | 1
Hyperhidrosis (General disorders) | 7
Influenza like illness (General disorders) | 2
Irritability (General disorders) | 3
Lethargy (General disorders) | 5
Oedema (General disorders) | 3
Oedema peripheral (General disorders) | 6
Pain (General disorders) | 9
Thirst (General disorders) | 1
Withdrawal syndrome (General disorders) | 1
Chronic hepatitis (Hepatobiliary disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Urticaria (Immune system disorders) | 4
Bronchitis (Infections and infestations) | 4
Candidiasis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 1
Localised infection (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 8
Oral candidiasis (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Pharyngitis streptococcal (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 3
Staphylococcal infection (Infections and infestations) | 1
Tooth infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 6
Urinary tract infection (Infections and infestations) | 2
Vulvovaginal mycotic infection (Infections and infestations) | 1
Accidental overdose (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 3
Fall (Injury, poisoning and procedural complications) | 1
Foot fracture (Injury, poisoning and procedural complications) | 1
Foreign body (Injury, poisoning and procedural complications) | 1
Hand fracture (Injury, poisoning and procedural complications) | 1
Joint injury (Injury, poisoning and procedural complications) | 1
Muscle strain (Injury, poisoning and procedural complications) | 1
Rotator cuff syndrome (Injury, poisoning and procedural complications) | 1
Skeletal injury (Injury, poisoning and procedural complications) | 1
Skin laceration (Injury, poisoning and procedural complications) | 1
Tendonitis (Injury, poisoning and procedural complications) | 1
Thermal burn (Injury, poisoning and procedural complications) | 1
Blood pressure increased (Investigations) | 1
Intraocular pressure increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 5
Dehydration (Metabolism and nutrition disorders) | 1
Gout (Metabolism and nutrition disorders) | 1
Obesity (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 6
Gout (Musculoskeletal and connective tissue disorders) | 2
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Restless legs syndrome (Musculoskeletal and connective tissue disorders) | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1
Abnormal dreams (Nervous system disorders) | 2
Agitation (Nervous system disorders) | 2
Balance disorder (Nervous system disorders) | 1
Carpal tunnel syndrome (Nervous system disorders) | 1
Cognitive disorder (Nervous system disorders) | 4
Confusional state (Nervous system disorders) | 5
Disorientation (Nervous system disorders) | 2
Disturbance in attention (Nervous system disorders) | 3
Dizziness (Nervous system disorders) | 17
Dysaesthesia (Nervous system disorders) | 1
Dysarthria (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Dysphemia (Nervous system disorders) | 1
Dysphonia (Nervous system disorders) | 2
Headache (Nervous system disorders) | 37
Hypoaesthesia (Nervous system disorders) | 1
Insomnia (Nervous system disorders) | 12
Paraesthesia (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Restless legs syndrome (Nervous system disorders) | 1
Restlessness (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 1
Sedation (Nervous system disorders) | 4
Sinus headache (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 25
Tension headache (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 4
Urinary incontinence (Nervous system disorders) | 1
Affective disorder (Psychiatric disorders) | 1
Aggression (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 2
Crying (Psychiatric disorders) | 1
Delirium (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 3
Dysphoria (Psychiatric disorders) | 1
Emotional disorder (Psychiatric disorders) | 1
Enuresis (Psychiatric disorders) | 1
Hallucination (Psychiatric disorders) | 2
Hallucinations, mixed (Psychiatric disorders) | 1
Hypersomnia (Psychiatric disorders) | 3
Mood swings (Psychiatric disorders) | 1
Nervousness (Psychiatric disorders) | 3
Nightmare (Psychiatric disorders) | 3
Throat tightness (Psychiatric disorders) | 1
Dysuria (Renal and urinary disorders) | 4
Pollakiuria (Renal and urinary disorders) | 1
Urinary hesitation (Renal and urinary disorders) | 2
Urinary retention (Renal and urinary disorders) | 2
Ejaculation disorder (Reproductive system and breast disorders) | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1
Hot flush (Reproductive system and breast disorders) | 1
Polymenorrhoea (Reproductive system and breast disorders) | 1
Sexual dysfunction (Reproductive system and breast disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2
Acne (Skin and subcutaneous tissue disorders) | 2
Night sweats (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 18
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 8
Rash generalised (Skin and subcutaneous tissue disorders) | 1
Swelling face (Skin and subcutaneous tissue disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
The study was prematurely terminated due to drug supply issues.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.